CLINICAL TRIAL: NCT03793179
Title: EA5163/S1709 INSIGNA : A Randomized, Phase III Study of Firstline Immunotherapy Alone or in Combination With Chemotherapy in Induction/Maintenance or Postprogression in Advanced Nonsquamous Non-Small Cell Lung Cancer (NSCLC) With Immunobiomarker SIGNature-Driven Analysis
Brief Title: Testing the Timing of Pembrolizumab Alone or With Chemotherapy as First Line Treatment and Maintenance in Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-03695; NCI-2018-03695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5163 (Other: ECOG-ACRIN Cancer Research Group); EA5163 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lung Non-Squamous Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; Carboplatin; Magnetic Resonance Spectroscopy; pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (pembrolizumab, pemetrexed, carboplatin) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Within 6 weeks of disease progression, patients receive pemetrexed IV over 10 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then may receive pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI during screening, CT scan and blood sample collection throughout the study, and may undergo PET scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Drug: Pemetrexed; Procedure: Positron Emission Tomography
- Arm B (pembrolizumab, pemetrexed, carboplatin) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Within 6 weeks of disease progression, patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pembrolizumab IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days for up to 2 years for pembrolizumab in the absence of disease progression or unacceptable toxicity and until to disease progression for pemetrexed. Patients undergo MRI during screening, CT scan and blood sample collection throughout the study, and may undergo PET scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Drug: Pemetrexed; Procedure: Positron Emission Tomography
- Arm C (pembrolizumab, pembrolizumab, carboplatin) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pembrolizumab IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days for up to 2 years for pembrolizumab in the absence of disease progression or unacceptable toxicity and until to disease progression for pemetrexed. Patients undergo MRI during screening, CT scan and blood sample collection throughout the study, and may undergo PET scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Drug: Pemetrexed; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase III trial studies whether pembrolizumab alone as a first-line treatment, followed by pemetrexed and carboplatin with or without pembrolizumab after disease progression is superior to induction with pembrolizumab, pemetrexed and carboplatin followed by pembrolizumab and pemetrexed maintenance in treating patients with stage IV non-squamous non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. It is not yet known whether giving first-line pembrolizumab followed by pemetrexed and carboplatin with or without pembrolizumab works better in treating patients with non-squamous non-small cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate overall survival (OS) in each of the 2 experimental arms (Arms A and B) to control (Arm C).

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for Arm C versus each of Arms A and B.

II. To evaluate best objective response rates per RECIST 1.1 for Arm C versus each of Arms A and B.

III. To estimate toxicity within each of the treatment arms via the Common Terminology Criteria for Adverse Events (CTCAE) criteria.

IV. To compare outcomes between Arms A and B. V. To compare outcomes by treatment arm within subgroups defined by a cutpoint of PD-L1 expression at >= 50%.

BIOMARKER OBJECTIVE:

I. To collect and bank tissue and blood for future research studies, including potential development of a prognostic and predictive signature for pembrolizumab (MK-3475) in combination with chemotherapy versus pembrolizumab (MK-3475) alone.

EXPLORATORY IMAGING OBJECTIVES:

I. To collect and bank standard of care computed tomography (CT) imaging at baseline and first three follow-up post-treatment scans on first line treatment for validating the radiomic risk score with the following exploratory objectives:

Ia. To determine the negative predictive value (NPV) by validating the Radiomic Risk score on pre-treatment scans as well as compute differences between pre- and post- treatment scans (delta features) in determining which patients will benefit from first line pembrolizumab in the metastatic setting in both low (< 50%) and high (> 50%) PD-L1 cohorts using patients in Arm 1 and Arm 2 of the trial where pembrolizumab is used as first line treatment.

Ib. To determine the positive predictive value (PPV) by validating the Radiomic Risk score in order to predict which patients would benefit from combination pembrolizumab and subsequent chemotherapy versus (vs.) immunotherapy alone in both low (< 50%) and high (> 50%) PD-L1 cohorts using patients who went on to receive chemotherapy as second line and stratifying the patients based on those who received benefit from pembrolizumab plus chemotherapy vs.pembrolizumab alone.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Within 6 weeks of disease progression, patients receive pemetrexed IV over 10 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then may receive pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Within 6 weeks of disease progression, patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pembrolizumab IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days for up to 2 years for pembrolizumab in the absence of disease progression or unacceptable toxicity and until to disease progression for pemetrexed.

ARM C: Patients receive pembrolizumab IV over 30 minutes, pemetrexed IV over 10 minutes, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive pembrolizumab IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days for up to 2 years for pembrolizumab in the absence of disease progression or unacceptable toxicity and until to disease progression for pemetrexed.

Patients undergo magnetic resonance imaging (MRI) during screening, CT scan and blood sample collection throughout the study, and may undergo position emission tomography (PET) scan throughout the study.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV non-squamous non-small cell lung cancer (NSCLC) (includes M1a, M1b, and M1c stage disease, American Joint Committee on Cancer [AJCC] 8th edition). Patients with stage IIIB and IIIC disease are eligible if they are not candidates for combined chemotherapy and radiation. Prior chemo-radiation therapy (RT) for stage III with recurrence is allowed
* Patients must have PD-L1 expression Tumor Proportion Score (TPS) >= 1% in tumor cells. If PD-L1 expression TPS is unevaluable or the testing could not be completed, the patients are not eligible. The assay must have been performed by a Clinical Laboratory Improvement Act (CLIA) (or equivalent) certified laboratory
* Patients must have measurable or non-measurable disease. The presence of malignant pleural fluid alone is sufficient to satisfy this eligibility criterion. Baseline imaging assessments and measurements used to evaluate all measurable or non-measurable sites of disease must be done within 4 weeks prior to study registration

  * NOTE: If patient receives pemetrexed, follow institutional guidelines to drain fluids
  * NOTE: An additional 15 days is allowed to account for any infection/exposure related logistical delays
* Patients must be >= 18 years of age
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Patients must NOT have received the following:

  * Prior systemic chemotherapy or immunotherapy for advanced metastatic NSCLC. Patients treated with any prior checkpoint inhibitors for metastatic lung cancer are ineligible. Chemotherapy for non-metastatic disease (e.g. adjuvant therapy) or immunotherapy for locally advanced stage III disease, or treated with neoadjuvant IO is allowed if at least 6 months have elapsed between the last dose of the prior therapy and study registration. Local therapy, e.g. palliative radiation, is allowed as long as a period of 14 days has passed between completion of local therapy and the start of protocol treatment. Registration during the 14 days is allowed. Palliative radiation must be to non-target lesions. Palliative radiation to pre-existing lesions while on protocol treatment is allowed as long as these areas have not grown to RECIST defined progression. Development of any new metastasis is considered progression. Concurrent radiation and protocol treatment is not allowed; protocol treatment may resume after completion of radiation as long as patient does not have greater than grade 2 side effects from radiation per physician discretion.
  * Methotrexate (MTX) given in low doses for non-malignant conditions with last dose at least 14 days prior to date of registration will be allowed. Other low dose chemotherapeutics for non-malignant conditions will be considered, but review by the study chair is required
  * Palliative radiation to non-target lesions (bone metastasis) is allowed if patient develops symptoms
* Patients with known EGFR mutations (except exon 20 insertion), BRAF mutations (V600) or ALK or ROS1 translocations or other driver mutations that can be treated with oral tyrosine kinase inhibitors are excluded
* Patients with treated brain metastases are eligible if follow-up brain imaging obtained at least 14 days after central nervous system (CNS)-directed therapy shows no evidence of progression. CNS progression counts as progression and patients must move on to the next phase after CNS treatment. Patients with asymptomatic new (at screening) or progressive brain metastases (active brain metastases at screening) are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy

  * Patients are eligible if off steroids for at least 14 days prior to protocol treatment
  * Anticonvulsants are allowed
  * Patients with asymptomatic, sub-centimeter brain metastasis who at the discretion of investigators do not need immediate CNS directed therapies are eligible
* Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients must not have known pre-existing and clinically active interstitial lung disease, or a known history of (non infectious) pneumonitis that required steroids, or current pneumonitis
* Patients must not have significant gastrointestinal disorders with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, etc.)
* Patients must not have history of auto-immune condition (including Guillain-Barre Syndrome or Multiple Sclerosis) requiring ongoing or intermittent systemic treatment in the past 2 years prior to registration (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must not have any other concomitant serious illness or organ system dysfunction that in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the study drug
* Patients must not receive any other investigational agents during the course of therapy
* Patients must not be pregnant or breast-feeding due to potential harm to the fetus or infant from cytotoxic chemotherapy and the unknown risk of pembrolizumab (MK-3475). All patients of childbearing potential must have a blood test or urine study within 72 hours prior to registration to rule out pregnancy. A patient of childbearing potential is someone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point; 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must use accepted and effective method(s) of contraception or by abstaining from sexual intercourse from time of registration, while on study treatment, and continue for 120 days after the last dose of study treatment
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within 14 days prior to randomization)
* Platelets >= 100,000/mm^3 (within 14 days prior to randomization)
* Prothrombin time (PT)/international normalized ratio (INR) (only if on active anticoagulation with warfarin or any formulations of heparin) =< 3.0 (within 14 day prior to randomization)
* Total bilirubin =< 1.5 mg/dL (obtained within 14 days prior to randomization)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) < 5 x upper limit of normal (ULN) (obtained within 14 days prior to randomization)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 5 x upper limit of normal (ULN) (obtained within 14 days prior to randomization)
* Calculated creatinine clearance >= 45 ml/min to be eligible to receive pemetrexed (obtained within 14 days prior to randomization)
* Serum creatinine =< 1.5 x institutional upper limit of normal (ULN) (obtained within 14 days prior to randomization)
* Patients must not have a known history of active tuberculosis (TB)
* Patients must not have a diagnosis of immunodeficiency or receive systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of protocol treatment
* Patients must not have received a live vaccine within 30 days prior to randomization. Patients are permitted to receive inactivated vaccines and any non-live vaccines including those for the seasonal influenza and COVID-19 (Note: intranasal influenza vaccines, such as Flu-Mist [registered trademark] are live attenuated vaccines and are not allowed). If possible, it is recommended to separate study drug administration from vaccine administration by about a week (primarily, in order to minimize an overlap of adverse events)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable or on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 5 years post treatment
  OS distributions will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to documented disease progression or death from any cause, assessed up to 5 years post treatment
  PFS distributions will be estimated using the Kaplan-Meier method.
Best objective response | Up to 5 years post treatment
  Best objective response will be evaluated via Response Evaluation Criteria in Solid Tumors 1.1 criteria.
Incidence of adverse events | Up to 30 days post treatment
  Toxicities will be reported via the Common Terminology Criteria for Adverse Events criteria version 5.0. Toxicity rates between arms in the overall population will be compared using Fisher's exact tests with a one-sided type I error rate of 1.25%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes.
PD-L1 positivity | At baseline
  PD-L1 positivity will be defined as >= 1% Tumor Proportion Score (TPS) for the purpose of enrollment onto the trial. Strongly PD-L1 positive is defined as >= 50% TPS; weakly positive is defined as 1% - 49% TPS.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Borghaei, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1097):
- United States (1084):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente Dublin, Dublin, California
  - 21st Century Oncology - El Segundo, El Segundo, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Aventura, Aventura, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - GenesisCare USA - Boca Raton FP02, Boca Raton, Florida
  - GenesisCare USA - Boca Ration FP06, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - GenesisCare USA - Gladiolus, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - GenesisCare USA - Key West, Key West, Florida
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - GenesisCare USA - Palm Beach Gardens, Palm Beach Gardens, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - The Longstreet Clinic - Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Freeman Physician Group of Pittsburg, Pittsburg, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - West Jefferson Medical Center, Marrero, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Veteran's Administration Medical Center - New Orleans, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Lourdes Hospital, Binghamton, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Levine Cancer Institute - Union West, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - WG Hefner VA Medical Center, Salisbury, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC Cancer Center-Bethel Park, Bethel Park, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Oncology Hematology Association, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University Cancer Specialists - Alcoa, Alcoa, Tennessee
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Tarrant County Hospital District/JPS Health Network, Fort Worth, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - SSM Health Dean Medical Group - Baraboo, Baraboo, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - SSM Health Dean Medical Group - Janesville, Janesville, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (12):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Niagara Health System-Saint Catharines General, Saint Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHA Hopital L'Enfant-Jesus, Québec, Quebec
- FHP Health Center-Guam, Tamuning, Guam

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT03793179/ICF_000.pdf